CLINICAL TRIAL: NCT06415994
Title: Multimodal Fetal and Placental Imaging and Biomarkers of Clinical Outcomes in Opioid Use Disorder
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rupa Radhakrishnan, Associate Professor of Radiology & Imaging Sciences, Indiana University
Other Study IDs: RADY-IIR-19751; R01DA059321 (NIH)
Record Dates: First submitted 2024-03-04; First posted 2024-05-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder; Substance-Related Disorders; Pregnancy Related; Narcotic-Related Disorders; Buprenorphine Dependence; Methadone Dependence
Keywords: Pregnant with Opioid Use Disorder; Opioid Use Disorder; Subutex; Buprenorphine; Pregnant taking buprenorphine/subutex
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Narcotic-Related Disorders | interventions — Buprenorphine; Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected at MRI visits for substances, DNA, RNA and epigenetic analysis.
  Placental sample: A sample of the placenta will be collected during delivery for analysis DNA, RNA and epigenetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant Mothers with Opioid Use Disorder: 150 pregnant mothers with opioid use disorder who are on buprenorphine or methadone treatment
  Interventions: Drug: Buprenorphine or Methadone Treatment; Diagnostic Test: Fetal and Placental MRI; Behavioral: Child Developmental Assessment; Behavioral: Questionnaires; Other: Blood and Placental Samples
- Pregnant Mothers: 100 pregnant mother who to not have a history of opioid use disorder
  Interventions: Diagnostic Test: Fetal and Placental MRI; Behavioral: Child Developmental Assessment; Behavioral: Questionnaires; Other: Blood and Placental Samples

INTERVENTIONS:
Drug: Buprenorphine or Methadone Treatment — Pregnant mothers must be taking Buprenorphine or Methadone
  Groups: Pregnant Mothers with Opioid Use Disorder
Diagnostic Test: Fetal and Placental MRI — Two MRIs :
  * Second Trimester
  * Third Trimester
Behavioral: Child Developmental Assessment — At 1 year of life child will receive a developmental assessment
Behavioral: Questionnaires — Participants will answer questionnaires on their medical history, pregnancy, substance use, and after birth: their child's development
Other: Blood and Placental Samples — At each MRI visit a blood sample will be collected for substances, DNA, RNA, epigenetics, and placental biomarkers.
  At delivery: A sample of placenta will be collected for RNA, DNA, and epigenetic analysis.

SUMMARY:
The goal of this observational study is to learn about the long term effects of prenatal opioid exposure. The main objectives are:

* Long term goal: to improve the safety and efficacy of maternal Opioid Use Disorder (OUD) and eliminate neonatal opioid withdrawal syndrome (NOWS) and poor childhood neurodevelopment.
* To characterize prenatal opioid exposure (POE) related placental and fetal brain structural and functional disruptions using longitudinal placenta-fetal brain magnetic resonance imaging (MRI) and determine proteomic, genomic, and epigenetic signatures of NOWS and poor infant neurodevelopment.

In this study participants will:

* Receive two placental-fetal MRIs, one during second trimester and one in third trimester.
* Answer surveys relating to their medical and social history.
* Have blood drawn during pregnancy and delivery.
* Child development follow up: answer surveys on their child's development milestones and at one year of life they will undergo a development assessment.

ELIGIBILITY:
Pregnant women with opioid use disorder

Inclusion Criteria:

* Age >18 years
* Currently taking buprenorphine or methadone for OUD and are enrolled in a prenatal opioid maintenance program
* Singleton Pregnancy
* Planned delivery at Indiana University or University of Pittsburgh study sites

Exclusion Criteria:

* Serious maternal medical illness as deemed by study physician investigators that would make it challenging to comply with study procedures
* Known or suspected major fetal/ neonatal congenital abnormalities
* HIV or AIDS

Infants with prenatal opioid exposure:

Inclusion:

1. Prenatal buprenorphine or methadone exposure
2. Born to mother enrolled in Opioid Use Disorder arm of study

Exclusion:

Major congenital anomalies or genetic syndromes affecting neurodevelopment

Control Pregnant Women:

Inclusion:

1. Women >18 Years of age
2. Healthy singleton pregnancy
3. Planned delivery at Indiana University or University of Pittsburgh study sites

Exclusion:

1. Serious maternal medical illness as deemed by study physician investigators that would make it challenging to comply with study procedures
2. HIV or AIDS
3. Known or suspected major fetal congenital abnormalities
4. Any history of opioid misuse before or during pregnancy-per self-report and clinical notes.

Control infants:

Inclusion:

Born to control pregnant mother enrolled in study

Exclusion:

Any major congenital anomalies, genetic abnormalities, neurologic abnormalities, syndromes, or chronic medical conditions affecting neurodevelopment.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any woman of the age of 18 or older that is having a single pregnancy, and currently taking buprenorphine or methadone for opioid use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Alterations in fetal brain volume | Between 20 weeks gestation and delivery
  Comparing changes in fetal brain volume using MRI between babies who have had prenatal opioid exposure (POE) and controls
Differences in placenta signal | Between 20 weeks gestation and delivery
  Comparing differences in placenta signal using MRI between the POE group and controls

SECONDARY OUTCOMES:
Placental epigenetic changes related to POE | Between 20 weeks gestation and delivery
  Compare placental DNA methylation in POE group and control group
Placental dysfunction biomarkers related to POE | Between 20 weeks gestation and delivery
  Compare concentrations of blood proteins in POE group vs controls
Neonatal Opioid Withdrawal Syndrome (NOWS) severity | After birth through one year of life
  Measuring NOWs severity in the POE group using eat sleep console scores
Length of Hospital Stay | After birth through one year of life
  Measuring NOWs severity in the POE group using length of hospital stay
Ages and Stages Questionnaire Scores during infancy | After birth through one year of life
  Comparing neurodevelopment of POE group and controls using the ages and stages questionnaire at multiple time points in baby's first year of life. This questionnaire assesses infants developmental level. Scores can identify whether child is below cutoff and needs professional intervention, close to cutoff and requires more developmental support and learning, or above cutoff and on track.
Neurocognitive and behavioral development assessment (Bayley-4) at one year of age | After birth through one year of life
  Comparing neurodevelopment of POE group and controls using the Bayley's 4 assessment at one year of age. This assessment is administered by professionals to identify development delays in children.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Pittsburg, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided